CLINICAL TRIAL: NCT02613143
Title: Zonulo-hyaloido-vitrectomy for Malignant Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: DXX-WZ
Record Dates: First submitted 2015-11-16; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Glaucoma
Keywords: malignant glaucoma; zonulo-hyaloido-vitrectomy

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Surgery

SUMMARY:
The purpose of this study is to assess the zonulo-hyaloido-vitrectomy for malignant glaucoma through an anterior approach.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent the zonulo-hyaloido-vitrectomy for malignant glaucoma through an anterior approach

Exclusion Criteria:

* systemic disease or inflammation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was consisted of patients who underwent the zonulo-hyaloido-vitrectomy for malignant glaucoma through an anterior approach. The Office of Research Ethics,Eye Hospital of Wenzhou Medical University approved the study protocol, and all patients provided their informed consent.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | 3 years
  The intraocular pressure is measured by the non-contact tonometer.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-e Zhao, MD, Study Chair — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China